CLINICAL TRIAL: NCT04374630
Title: An Open Label Randomized Active Controlled Phase II Clinical Study to Assess the Efficacy and Safety of Afuresertib Plus Paclitaxel Versus Paclitaxel in Patients With Platinum-Resistant Ovarian Cancer
Brief Title: Study With Afuresertib and Paclitaxel in Platinum Resistant Ovarian
Acronym: PROFECTA-II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laekna Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAE002INT2001
Record Dates: First submitted 2020-04-02; First posted 2020-05-05 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-03

CONDITIONS: Platinum-resistant Ovarian Cancer
MeSH Terms: interventions — Paclitaxel; afuresertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Arm 1 is afuresertib 125 mg PO QD + paclitaxel 80 mg/m2 intravenous (IV) infusion over 1 hour on Days 1, 8 and 15 of a 3 week cycle.
  Interventions: Drug: Paclitaxel; Drug: Afuresertib
- Arm 2 (Active Comparator): Arm 2 is paclitaxel 80 mg/m2 IV infusion over 1 hour on Days 1, 8, and 15 of a 3 week cycle
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Commercially available paclitaxel for IV administration will be obtained by clinical sites in US.
Drug: Afuresertib — Each afuresertib 50 mg tablet, intended for oral administration, contains afuresertib (hydrochloride salt) equivalent to 50 mg of afuresertib (free base).
  Each afuresertib 75 mg tablet, intended for oral administration, contains afuresertib (hydrochloride salt) equivalent to 75 mg of afuresertib (free base)
  Other Names: LAE002
  Arms: Arm 1

SUMMARY:
Afuresertib is an AKT inhibitor, a new class of agents under development that may provide physicians with a new clinical option to control platinum resistant ovarian cancer (PROC) progression. Afuresertib plus chemotherapy has demonstrated anti-tumor efficacy and an acceptable safety profile in patients with PROC in a published Phase I/II study. Therefore, the combination of afuresertib plus weekly paclitaxel could represent a clinically meaningful step forward in the clinical management of these difficult-to-treat patients with PROC.

DETAILED DESCRIPTION:
A total of approximately 141 patients with PROC are planned to be enrolled and randomized with a 2:1 ratio in an open label manner to the 2 arms (94 patients in the combination treatment arm and 47 patients in the paclitaxel arm) for efficacy and safety evaluation. The randomization will be stratified by country (the United States vs. China), prior bevacizumab use (yes vs. no), and number of prior platinum based therapy treatments (1-2 vs. 3-5 prior platinum regimens). The study will consist of 3 periods. The first period is the Screening Period (Day -24 to 1) during which patients are screened for eligibility according to the inclusion and exclusion criteria. The second period is a Treatment Evaluation Period with a randomized, open-label, two arm parallel design (from starting study treatment until patients have progressive disease [PD], unacceptable toxicity, death, or withdrawal of consent). The PK study will be applied to both the combination treatment arm and control arm. The third period is a Follow up Period (safety evaluation at 30 days after the last dose of study treatment and OS and/or PFS follow up). Patients will be tested at baseline for phosphoinositide 3 kinase (PI3K)/AKT/PTEN pathway alterations and BRCA1/2 mutations by NGS, and/or level of phospho AKT by IHC; the correlation of the efficacy endpoints and biomarker status will be analyzed retrospectively as an exploratory endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. 1. Female patients at least 18 years of age at the time of signing the informed consent form and capable of giving written informed consent, which includes willingness to comply with the requirements and restrictions listed in the consent form.
2. Must provide informed consent for the procedures and the tests for PI3K/AKT/PTEN pathway alterations, BRCA1/2 mutations, and/or level of phospho-AKT. The archival tumor biopsy sample collected less than 1 year is preferred. If no archival tumor sample is available, fresh biopsy will be recommended. For patients who cannot provide a tumor sample or cannot accept fresh tumor biopsy, the Sponsor should be consulted about their qualification to enter this study.
3. Patients must have histologically or cytologically confirmed high grade serous OC, endometroid OC, or ovarian clear cell carcinoma (including fallopian tube and primary peritoneal cancers). Carcinosarcoma, sarcoma, mucinous OC, or low-grade serous OC or the other histologies must be excluded.
4. Must not have previously received prior AKT or PI3K pathway or mTOR inhibitors.
5. Must have PROC (including fallopian tube and primary peritoneal carcinoma), defined as disease relapsed between 1 to 6 months after the last dose of the first-line platinum-based therapy (at least 3 cycles), or progressed during or relapsed within 6 months of the last dose of platinum-based 2nd-5th line therapies.
6. The OC patients must have received 1 to 5 prior chemotherapies including no more than one chemotherapy after PROC was diagnosed. Combination therapy with two or more drugs will be considered as one therapy, whereas maintenance therapy will be considered as continuation of the previous systemic treatment.
7. Patients should be appropriate candidates for treatment with single agent weekly paclitaxel based on investigator's clinical assessment.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
9. Must meet the following criteria for hematology parameters:

   * Absolute neutrophil count (ANC) ≥ 1,500/mm3
   * Platelets ≥ 100,000/µL
   * Hemoglobin ≥ 9.0 g/dL
10. Total serum bilirubin ≤ 1.5 × upper limit of normal (ULN) (in patients with known Gilbert's syndrome, total bilirubin ≤ 3 × ULN with direct bilirubin ≤ 1.5 × ULN).
11. Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) must be < 2.5 × institutional ULN. For patients with liver metastasis, AST/ALT must be < 5.0 × institutional ULN.
12. Creatinine within 1.5 × ULN or creatinine clearance > 30 mL/min by Cockcroft Gault formula (Appendix 1).
13. Toxicities of prior therapy (except alopecia) should have been resolved to less than or equal to grade 1 as per NCI-CTCAE v5.0.
14. Patients must have GI functions that would allow absorption of afuresertib.
15. Patient must have a life expectancy of greater than 6 months.
16. Must have at least one lesion that meets the definition of measurable disease by RECIST 1.1 criteria (Appendix 3).
17. Patients of childbearing potential must agree to use adequate contraception (barrier method of birth control or abstinence) prior to study entry and for the duration of study participation. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she should inform her treating physician immediately.
18. Must be off strong inhibitors or inducers of CYP3A4/5 treatment, as showed in Appendix 2, for at least 2 weeks from Study Day 1.

Exclusion Criteria:

1. 1. Primary platinum refractory disease, defined as "disease progression during or relapsed within 1 month after the last dose of the first-line platinum based therapy".
2. Known or suspected brain metastases.
3. Receiving any other anticancer therapeutic agents other than study medicines.
4. Uncontrolled ascites.
5. Known symptomatic or impending cord compression, except if the patient has received definitive treatment for this and demonstrates evidence of clinically stable disease.
6. Presence of other active cancer within 3 years prior to enrollment (other than basal cell or squamous cell skin cancer, or any other cancer in situ currently in complete remission).
7. History of seizure or condition that may predispose to seizure that needs anti-epileptic medications; brain arteriovenous malformation; or intracranial masses, such as schwannomas and meningiomas that are causing edema or mass effect.
8. Known allergies, hypersensitivity, or intolerance to the excipients of afuresertib (for excipient information, refer to the IB17).
9. Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the patient (eg, compromise well-being) or that could prevent, limit, or confound the protocol-specified assessments.
10. Any medical contraindication to the use of paclitaxel.
11. Prior radiotherapy ≤ 15 days prior to Study Day 1, with the exception of a single fraction of radiotherapy for the purposes of palliation, which is permitted.
12. History of clinically significant ventricular arrhythmias (eg, ventricular tachycardia, ventricular fibrillation, or torsade de pointes).
13. Prolonged corrected QT interval by the Fridericia's correction formula (QTcF) on the screening ECG > 470 msec. Receiving concomitant medications known to prolong QTc, or which are associated with torsade de pointes, and are unable to discontinue use while receiving study drug.
14. History or evidence for any of the following: severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (eg, pulmonary embolism, cerebrovascular accident including transient ischemic attacks) within 6 months prior to Study Day 1 or New York Heart Association Class III to IV heart disease.
15. Presence of uncontrolled hypertension (systolic blood pressure [BP] > 160 mmHg or diastolic BP > 100 mmHg). Patients with a history of hypertension are allowed, provided that BP is controlled to within these limits by anti-hypertensive treatment.
16. Human immunodeficiency virus (HIV)-positive patients with 1 or more of the following:

    1. Not receiving highly active antiretroviral therapy
    2. Receiving antiretroviral therapy that may interfere with the study drug (consult the Sponsor for review of medication prior to enrollment)
    3. CD4 count < 350 based on a test within 3 months of the screening visit
    4. An acquired immunodeficiency syndrome-defining opportunistic infection within 6 months of the start of screening
17. Had a major surgery ≤ 30 days prior to first study treatment at Cycle 1 Day 1.
18. Presence of grade > 2 neuropathy.
19. Prior receipt of chemotherapy, PARP inhibitor, bevacizumab, or investigational therapy within 28 days of enrollment or within 5 half lives of the agent, whichever is shorter.
20. Patients who are pregnant or lactating.
21. Patients with high risk of tuberculosis infection, based on investigator's clinical assessment, will be screened by tuberculosis screening test, such as the QuantiFERON® TB Gold In Tube test (QFT-GIT) or the T-SPOT®.TB test (T-Spot).
22. Patients with active hepatitis B (positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C (positive hepatitis C virus [HCV] antibody test at screening) are not allowed to be enrolled in this study. Note:

    * Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive hepatitis B core antibody [HBcAb] test) are eligible.
    * Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
PFS based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Change from Baseline every 6 weeks × 30 weeks, then every 8 weeks through study completion, an average of 1 year
  Radiographic imaging will be performed and assessed by investigators

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization until date of death, from any cause, assessed up to 1 year.
  To further evaluate the clinical efficacy via OS collection
Objective response rate (ORR) according to RECIST 1.1 | Change from Baseline every 6 weeks × 30 weeks, then every 8 weeks through study completion, an average 1 year.
  To further evaluate the clinical efficacy via ORR
Duration of response (DOR) according to RECIST 1.1 | Change from Baseline every 6 weeks × 30 weeks, then every 8 weeks through study completion, an average of 1 year.
  To further evaluate the clinical efficacy via DOR
Disease control rate (DCR) according to RECIST 1.1 | Change from Baseline every 6 weeks × 30 weeks, then every 8 weeks through study completion, an average of 1 year.
  To further evaluate the clinical efficacy via DCR
Best overall response (BOR) according to RECIST 1.1 | Change form Baseline every 6 weeks × 30 weeks, then every 8 weeks through study completion, an average of 1 year.
  To further evaluate the clinical efficacy via BOR
Cancer antigen 125 (CA-125) response (Gynecological Cancer Intergroup [GCIG]) | Change from Baseline every 6 weeks × 30 weeks, then every 8 weeks through study completion, an average of 1 year.
  To further evaluate the clinical efficacy via CA125 response
Area under the curve in the inter-dose interval period after first dose (AUCτ) | Samples collected on Cycle1Day1, Cycle2Day1, Cycle3Day1 and Cycle4Day1 will be assessed (a Cycle is 21 days)
  To Characterize Pharmacokinetics (PK) of afuresertib and paclitaxel in patients with PROC under combination therapy of afuresertib plus paclitaxel, or paclitaxel alone at steady-state via AUCτ
Area under the curve in the inter-dose interval period at steady state (AUCτ_SS) | Samples collected on Cycle1Day1, Cycle2Day1, Cycle3Day1 and Cycle4Day1 will be assessed (a Cycle is 21 days)
  To Characterize Pharmacokinetics (PK) of afuresertib and paclitaxel in patients with PROC under combination therapy of afuresertib plus paclitaxel, or paclitaxel alone at steady-state via AUCτ_SS
Maximum concentration after first dose (Cmax) | Samples collected on Cycle1Day1, Cycle2Day1, Cycle3Day1 and Cycle4Day1 will be assessed (a Cycle is 21 days)
  To Characterize Pharmacokinetics (PK) of afuresertib and paclitaxel in patients with PROC under combination therapy of afuresertib plus paclitaxel, or paclitaxel alone at steady-state via Cmax
Maximum concentration at steady state (Cmax_SS) | Samples collected on Cycle1Day1, Cycle2Day1, Cycle3Day1 and Cycle4Day1 will be assessed (a Cycle is 21 days)
  To Characterize Pharmacokinetics (PK) of afuresertib and paclitaxel in patients with PROC under combination therapy of afuresertib plus paclitaxel, or paclitaxel alone at steady-state via Cmax_SS
Time to maximum concentration after first dose (Tmax) To explore potential effect of coadministration of afuresertib | Samples collected on Cycle1Day1, Cycle2Day1, Cycle3Day1 and Cycle4Day1 will be assessed(a Cycle is 21 days)
  To Characterize Pharmacokinetics (PK) of afuresertib and paclitaxel in patients with PROC under combination therapy of afuresertib plus paclitaxel, or paclitaxel alone at steady-state via Tmax
Time to maximum concentration at steady state (Tmax_SS) | Samples collected on Cycle1Day1, Cycle2Day1, Cycle3Day1 and Cycle4Day1 will be assessed (a Cycle is 21 days)
  To Characterize Pharmacokinetics (PK) of afuresertib and paclitaxel in patients with PROC under combination therapy of afuresertib plus paclitaxel, or paclitaxel alone at steady-state via Tmax_SS
Half-life (T1/2) if data permit | Samples collected on Cycle1Day1, Cycle2Day1, Cycle3Day1 and Cycle4Day1 will be assessed(a Cycle is 21 days)
  To Characterize Pharmacokinetics (PK) of afuresertib and paclitaxel in patients with PROC under combination therapy of afuresertib plus paclitaxel, or paclitaxel alone at steady-state via T1/2
Trough concentration at steady state (Ctrough_SS) | Samples collected on Cycle1Day1, Cycle2Day1, Cycle3Day1 and Cycle4Day1 will be assessed (a Cycle is 21 days)
  To Characterize Pharmacokinetics (PK) of afuresertib and paclitaxel in patients with PROC under combination therapy of afuresertib plus paclitaxel, or paclitaxel alone at steady state via Ctrough_SS
Rate and severity of treatment-emergent adverse events (TEAEs) based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 | From date of consent until 30 days following discontinuation of study treatment
  Patients to be queried as to whether they have experienced adverse event
Vital signs-Blood Pressure | Cycle1Day 1 and Cyle 1 D15, then on Day 1 of subsequent cycles
  Assessment of Blood Pressure
Vital signs-Heart Rate | Cycle1Day 1 and Cyle 1 D15, then on Day 1 of subsequent cycles
  Assessment of heart rate
Vital signs-Respiratory rate | Cycle1Day 1 and Cyle 1 D15, then on Day 1 of subsequent cycles
  Assessment of respiratory rate
Vital signs-body temperature | Cycle1Day 1 and Cyle 1 D15, then on Day 1 of subsequent cycles
  Assessment of body temperature.
Electrocardiogram (ECG) | Screening and repeated if clinically indicated through study completion, an average of 1 year.
  ECG QT Interval
Physical examinations | Assessment to be complete every 2 weeks for first 2 cycles, then once per cycle (each Cycle is 21 days)
  Assessment of head, eyes, ears, nose, and throat, chest, cardiac, abdominal, extremities, neurologic, and lymph node examinations
CBC | Screening then Cycles1 and 2 Day 1, 8,and 15 and D1 of subsequent cycles through study completion, an average up to 1 year.
  Assessment includes Platelet Count, Hemoglobin, WBC Count (absolute), Neutrophils, Lymphocytes, Eosinophils, Monocytes, Basophils
Clinical Chemistry | Screening and Day1 of each cycle through study completion, an avergae up to 1 year.
  Assessment includes BUN, Creatinine, Glucose (fasting), Sodium, Total Protein, Magnesium , Potassium, Chloride, Total CO2, Calcium, Albumin, AST (SGOT), ALT (SGPT), Phosphorous, Alkaline phosphatase, Total and direct bilirubin

OTHER OUTCOMES:
PFS based on RECIST 1.1 | After C2 (each cycle is 21 days), then every 6 weeks for 30 weeks, then every 8 weeks through study completion, an average up to 1 year.
  explore the PFS of the combination treatment arm versus paclitaxel arm in association with the biomarkers:
  * Alterations of PI3K/AKT/PTEN pathway and BRCA1/2 mutations in tumor samples as ssessed by next generation sequencing (NGS)
  * Levels of phospho-AKT in tumor sample as assessed by immunohistochemistry (IHC)
OS | From date of randomization until date of death
  explore the OS of the combination treatment arm versus paclitaxel arm in association with the biomarkers:
  * Alterations of PI3K/AKT/PTEN pathway and BRCA1/2 mutations in tumor samples as ssessed by next generation sequencing (NGS)
  * Levels of phospho-AKT in tumor sample as assessed by immunohistochemistry (IHC)
ORR based on RECIST 1.1 | After C2 (each cycle is 21 days), every 6 weeks x 30 weeks, then every 8 weeks through study completion, an avergae of 1 year.
  explore the ORR of the combination treatment arm versus paclitaxel arm in association with the biomarkers:
  * Alterations of PI3K/AKT/PTEN pathway and BRCA1/2 mutations in tumor samples as ssessed by next generation sequencing (NGS)
  * Levels of phospho-AKT in tumor sample as assessed by immunohistochemistry (IHC)
BOR based on RECIST 1.1 | After C2 (each cycle is 21 days), every 6 weeks x 30 weeks, then every 8 weeks through study completion, an avergae of 1 year.
  explore the BOR of the combination treatment arm versus paclitaxel arm in association with the biomarkers:
  * Alterations of PI3K/AKT/PTEN pathway and BRCA1/2 mutations in tumor samples as ssessed by next generation sequencing (NGS)
  * Levels of phospho-AKT in tumor sample as assessed by immunohistochemistry (IHC)
DOR based on RECIST 1.1 | After C2 (each cycle is 21 days), every 6 weeks x 30 weeks, then every 8 weeks through study completion, an average of 1 year.
  explore the DOR of the combination treatment arm versus paclitaxel arm in association with the biomarkers:
  * Alterations of PI3K/AKT/PTEN pathway and BRCA1/2 mutations in tumor samples as ssessed by next generation sequencing (NGS)
  * Levels of phospho-AKT in tumor sample as assessed by immunohistochemistry (IHC)
DCR based on RECIST 1.1 o Alterations of PI3K/AKT/PTEN pathway and BRCA1/2 mutations in tumor samples as assessed by next generation sequencing (NGS) o Levels of phospho AKT in tumor sample as assessed by immunohistochemistry (IHC) | After C2 (each cycle is 21 days), every 6 weeks x 30 weeks, then every 8 weeks through study completion, an avergae of 1 year.
  explore the DCR of the combination treatment arm versus paclitaxel arm in association with the biomarkers:
  * Alterations of PI3K/AKT/PTEN pathway and BRCA1/2 mutations in tumor samples as ssessed by next generation sequencing (NGS)
  * Levels of phospho-AKT in tumor sample as assessed by immunohistochemistry (IHC)
CA-125 response (GCIG) | Change from Baseline every 6 weeks × 30 weeks, then every 8 weeks through study completion, an averge of 1 year.
  explore the CA125 response of the combination treatment arm versus paclitaxel arm in association with the biomarkers:
  * Alterations of PI3K/AKT/PTEN pathway and BRCA1/2 mutations in tumor samples as ssessed by next generation sequencing (NGS)
  * Levels of phospho-AKT in tumor sample as assessed by immunohistochemistry (IHC)

CONTACTS AND LOCATIONS:
Overall Officials: Herzog Thomas, Professor, Principal Investigator — University of Cincinnati Medical Center/USA/1010
Locations (47):
- United States (30):
  - Arizona Oncology Associates, Phoenix, Arizona
  - Arizona Oncology, Tucson, Arizona
  - Highlands Oncology Group, Rogers, Arkansas
  - Gynecology Oncology Associates Newport Beach, Newport Beach, California
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - University of Chicago, Chicago, Illinois
  - Women's Cancer Care, Covington, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - MD Anderson Cancer Center at Cooper, Camden, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Southwest Women's Oncology Group, Albuquerque, New Mexico
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - OHCare Oncology Hematology Care (OHC), Inc. - Kenwood Office, Cincinnati, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Abington Memorial Hospital, Willow Grove, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - Texas Oncology, Austin, Texas
  - Texas Oncology, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - USO Texas Oncology, Longview, Texas
  - US Texas Oncology, San Antonio, Texas
  - Baylor Scott & White Medical Center, Temple, Texas
  - Texas Oncology, The Woodlands, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - University of Washington/Seattle Cancer Care Alliance, Seattle, Washington
- China (17):
  - Beijing Obstetrics & Gynecology Hospital, Capital Medical University, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Peking University Cancer Hospital, Beijing
  - Chongqing University Cancer Hospital, Chongqing
  - Sun Yat-sen University Cancer Center, Guangdong
  - Harbin Medical University Cancer Hospital, Heilongjiang
  - Henan Cancer Hospital, Henan
  - Hubei Cancer Hospital, Hubei
  - Hunan Cancer Hospital, Hunan
  - Jilin Cancer Hospital, Jilin
  - Liaoning Cancer Hospital, Liaoyang
  - Qilu Hospital of Shandong University, Shandong
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai
  - Zhongshan Hospital affiliated to Fudan University, Shanghai
  - West China Second University Hospital,Sichuan University, Sichuan
  - The Second Hospital of Tianjin Medical University, Tianjin
  - Women's Hospital school of medicine Zhejiang University, Zhejiang